CLINICAL TRIAL: NCT04039477
Title: A Phase 2 Randomized, Dose-blind, Multicenter Study to Evaluate the Safety and Efficacy of KZR-616 in the Treatment of Patients With Autoimmune Hemolytic Anemia (AIHA) and Immune Thrombocytopenia (ITP)
Brief Title: A Phase 2 Study to Evaluate the Safety and Efficacy of KZR-616 in Patients With AIHA and ITP
Acronym: MARINA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Clinical trial activity slowdown due to COVID-19 pandemic, high screen fail rate, and lack of enrollment led to the decision to withdraw the MARINA study.
Sponsor: Kezar Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KZR-616-005
Record Dates: First submitted 2019-07-26; First posted 2019-07-31 (Actual); Last update posted 2020-08-07 (Actual); Status verified 2020-08

CONDITIONS: Autoimmune Hemolytic Anemia; Immune Thrombocytopenia
Keywords: Autoimmune; Hemolytic; Anemia; Autoimmune Hemolytic Anemia; AIHA; Immune; Thrombocytopenia; Immune Thrombocytopenia; ITP; Blood disorders; Hematology
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune; Purpura, Thrombocytopenic, Idiopathic; Hemolysis; Anemia; Thrombocytopenia; Hematologic Diseases | interventions — KZR-616

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A - KZR-616 30mg (Experimental): KZR-616 30mg Subcutaneous (SC) injection weekly for 13 weeks
  Interventions: Drug: KZR-616
- Arm B - KZR-616 45mg (Experimental): KZR-616 30 mg SC injection weekly for 1 dose then 45mg weekly for 12 weeks.
  Interventions: Drug: KZR-616

INTERVENTIONS:
Drug: KZR-616 — Patients will receive KZR-616 SC once weekly. Patients assigned to Arm A will receive 30 mg for 13 weeks and patients assigned to Arm B will receive 30 mg for 1 week then 45 mg for 12 weeks

SUMMARY:
This is a Phase 2 randomized, dose-blind, multicenter study designed to evaluate the safety, tolerability, efficacy, Pharmacokinetics (PK), and Pharmacodynamics (PD) of treatment with KZR-616 in patients with active Autoimmune Hemolytic Anemia or Immune Thrombocytopenia.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients must be at least 18 years of age at the time of signing informed consent at Screening
2. Body Mass Index (BMI) equal to or greater than 18 kg/m2
3. Have a documented diagnosis of primary or secondary AIHA, ITP, or primary Evans syndrome
4. AIHA or ITP disease activity as follows::

   1. ITP: Per central or local laboratory assessments on 2 separate occasions ≥7 days apart during Screening, a mean Platelet (PLT) ≤30×109/L with no individual PLT >35×109/L; or for those patients receiving a constant dose of permitted treatments for ITP: a mean PLT <50×109/L, with no count >55×109/L
   2. AIHA: Hgb ≤10 g/dL and presence of any 2 of the following:

   i. Haptoglobin <lower limit of normal (LLN) ii. Corrected reticulocyte count >upper limit of normal (ULN) iii. LDH >ULN iv. Indirect bilirubin >ULN.
5. Documented inadequate response on intolerance to ≥1 standard treatment approach for AIHA or ≥2 standard treatment approaches for ITP

Exclusion Criteria:

1. Systemic Lupus Erythematosus (SLE) with confirmed anti-phospholipid antibody syndrome, the presence of positive lupus anti-coagulant test, moderate-high titer anti-cardiolipin IgG or IgM or moderate-high titer anti-beta2-globuilin IgG or IgM or severe central nervous system involvement
2. History of clinically significant coagulopathy, hereditary thrombocytopenia, anemia, or family history of thrombocytopenia
3. History of primary immunodeficiency
4. Use of nonpermitted medications within the specified washout periods prior to screening
5. Recent serious or ongoing infection, or risk for serious infection
6. Any of the following laboratory values at Screening:

   1. Estimated glomerular filtration rate (eGFR) <45 ml/min
   2. Absolute neutrophil count (ANC) <1.5×109/L (1500/mm3)
   3. Serum aspartate transaminase (AST), serum alanine transaminase (ALT) or serum alkaline phosphatase >2.5×ULN
   4. Thyroid stimulating hormone if outside of the central laboratory normal range and considered clinically significant
   5. International normalized ratio (INR) or activated partial thromboplastin time (aPTT) >1.5×ULN
   6. Immunoglobulin G (IgG) <500 mg/dL
   7. For ITP patients only: total bilirubin >1.5×ULN (3×ULN for patients with documented Gilbert's syndrome).
7. Presence of New York Heart Association Class III or IV heart failure, or uncontrolled blood pressure, or prolonged QT interval
8. Major surgery within 12 weeks before Screening or planned during the study period
9. History of any thrombotic or embolic event within 12 months prior to Screening
10. Clinical evidence of significant unstable or uncontrolled diseases
11. Any active or suspected malignancy or history of documented malignancy within the last 5 years before Screening, except appropriately excised and cured cervical carcinoma in situ or basal or squamous cell carcinoma of the skin, or non-muscle invasive bladder cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-07 (Estimated); Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Mean change from Baseline to Week 13 in hematologic parameters of interest in evaluable patients (Hgb for AIHA; Platelets [PLT] for ITP) | 13 weeks

SECONDARY OUTCOMES:
Mean change from Baseline to Week 13 in hematologic parameters of interest (Hgb for AIHA; PLT for ITP) in the intent to treat (ITT) population | 13 weeks
Mean change from Baseline over time in hematologic parameters of interest (Hgb for AIHA; PLT for ITP) | Through study completion, up to 25 weeks
Proportion of patients with a response at Week 13 | 13 weeks
Proportion of patients over time with a response | Through study completion, up to 25 weeks
Time to response | Through study completion, up to 25 weeks
Proportion of patients over time with loss of response | Through study completion, up to 25 weeks
Proportion of patients over time with sustained response | Through study completion, up to 25 weeks
Mean change from Baseline over time in Hct | Through study completion, up to 25 weeks
Mean change from Baseline over time in Lactate Dehydrogenase (LDH) | Through study completion, up to 25 weeks
Change from Baseline over time in Patient Global Assessment scores | Baseline and every 4 weeks for 25 weeks
  The PtGA is a visual analog scale (VAS) ranging from 0 to 100. Patients will provide a global rating of their disease, for the day of the visit, in response to the statement "Considering all the ways that your disease affects you, please rate how you are feeling today by clicking or tapping on the line:" using a 100-point VAS where 0 is "very good, no symptoms" and 100 is "very poor, very severe symptoms."
For AIHA: Proportion of patients with an Hgb >12 g/dL or 2 g/dL higher than Baseline at W13 | 13 weeks
For AIHA: Number of blood transfusions and units of blood administered over time | Through study completion, up to 25 weeks
For ITP: Number of platelet transfusions and units of platelets administered over time | Through study completion, up to 25 weeks
Safety and tolerability of KZR-616 in patients with AIHA or ITP as assessed by monitoring incidence and severity of adverse events (AEs) | Through study completion, up to 25 weeks
Peak Plasma Concentration (Cmax) following KZR-616 injection | Day 1
Peak Plasma Concentration (Cmax) following KZR-616 injection | Day 29
Time to peak plasma concentration (Tmax) following KZR-616 injection | Day 1
Time to peak plasma concentration (Tmax) following KZR-616 injection | Day 29
Area under the plasma concentration versus time curve (AUC) following KZR-616 injection | Day 1
Area under the plasma concentration versus time curve (AUC) following KZR-616 injection | Day 29
Half-life (T1/2) following KZR-616 injection | Day 1
Half-life (T1/2) following KZR-616 injection | Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Kezar, Study Director — Kezar Life Sciences, Inc.
Locations (22):
- United States (15):
  - KZR Research Site, Los Angeles, California
  - KZR Research Site, San Francisco, California
  - KZR Research Site, Jacksonville, Florida
  - KZR Research Site, Miami Lakes, Florida
  - KZR Research Site, Tampa, Florida
  - KZR Research Site, Peoria, Illinois
  - KZR Research Site, Boston, Massachusetts
  - KZR Research Site, Minneapolis, Minnesota
  - KZR-616 Research Site, Rochester, Minnesota
  - KZR Research Site, Morristown, New Jersey
  - KZR Research Site, The Bronx, New York
  - KZR Research Site, Greenville, North Carolina
  - KZR Research Site, Cleveland, Ohio
  - KZR Research Site, Columbus, Ohio
  - KZR Research Site, Webster, Texas
- KZR Research Site, Woolloongabba, Australia
- Italy (2):
  - KZR Research Site, Bologna
  - KZR Research Site, Genova
- Poland (2):
  - KZR Research Site, Krakow
  - KZR Research Site, Poznan
- Russia (2):
  - KZR Research Site, Moscow
  - KZR Research Site, Saint Petersburg

IPD SHARING:
Plan to Share IPD: No